CLINICAL TRIAL: NCT01621854
Title: A Two-part, Phase I Open Label Dose-escalation Study to Assess the Safety, Pharmacokinetics and Clinical Activity of NUC-1031, a Nucleotide Analogue, in Patients With Advanced Solid Tumours.
Brief Title: NUC-1031 in Patients With Advanced Solid Tumours
Acronym: ProGem1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Nucana (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-001
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cancer
Keywords: cancer; nucleoside analogue; advanced solid tumours
MeSH Terms: conditions — Neoplasms | interventions — NUC-1031

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NUC-1031 (Experimental): Cohort 1, Schedule A, NUC-1031 I.V. 1000mg/m2, Days 1, 8, & 15 every 28 days Cohort 1, Schedule B, NUC-1031 I.V. 500mg/m2, Days 1 & 5, 8 & 12, 15 &19 every 28 days Cohort 2, Schedule A, NUC-1031 I.V. 2000mg/m2, Days 1, 8, & 15 every 28 days Cohort 2, Schedule B, NUC-1031 I.V. 1000mg/m2, Days 1 & 5, 8 & 12, 15 &19 every 28 days
  Interventions: Drug: NUC-1031

INTERVENTIONS:
Drug: NUC-1031 — Cohort 1, Schedule A, NUC-1031 I.V. 1000mg/m2, Days 1, 8, & 15 every 28 days Cohort 1, Schedule B, NUC-1031 I.V. 500mg/m2, Days 1 & 5, 8 & 12, 15 &19 every 28 days Cohort 2, Schedule A, NUC-1031 I.V. 2000mg/m2, Days 1, 8, & 15 every 28 days Cohort 2, Schedule B, NUC-1031 I.V. 1000mg/m2, Days 1 & 5, 8 & 12, 15 &19 every 28 days

SUMMARY:
This is a two-part Phase I, open label, dose-escalation, study of NUC-1031 as a single agent in patients with advanced solid tumours who have failed to respond to or who have relapsed after treatment with standard therapy. NUC-1031 is a ProTide of gemcitabine, a drug that has been used widely and effectively against cancers for many years. Both NUC-1031 and gemcitabine work by preventing cancer cells from dividing by attacking their DNA (deoxyribonucleic acid). Non clinical studies have shown that NUC-1031 is more effective than gemcitabine because it is able to reach cancer cells by passive diffusion, is less easily degraded by the cancer cell, and delivers the monophosphate form of the active agent. The first part of the study is to determine recommended phase 2 dose by dose escalation and the second part is to explore preliminary anti-tumour activity.

DETAILED DESCRIPTION:
This is a two-part, Phase I, open label study of NUC-1031 as a single agent, administered IV weekly on days 1, 8, & 15 (Schedule A) or twice weekly on days 1 & 5, 8 & 12, 15 &19 (Schedule B) of a 28 day- cycle regimen. An initial dose-escalation phase (Part I) will be followed by an expansion cohort phase (Part II) using the preferred regimen from Part I. In Part I, sequential patients will be assigned to increasing doses of NUC-1031 in a standard '3 + 3' design to determine the recommended Phase II dose (RP2D). There will be a review of all available data (in particular the safety profile and preliminary PK data through to at least the last scheduled day of Cycle 1) following enrolment of the second cohort of both schedule A and B to select the preferred administration schedule to take forward for ongoing evaluation.

In Part II (dose expansion) additional patients will be enrolled to receive NUC-1031 at the RP2D and dosing frequency determined from Part I of the study. During Part II, further information will be obtained regarding safety, PK, PD and preliminary anti-tumour efficacy of NUC-1031 at RP2D.

In both parts of the study, patients may continue to receive NUC-1031 for up to 6 cycles, until disease progression, for as long as the participant receives clinical benefit in the opinion of the CI, the occurrence of unmanageable drug related toxicity despite dose modification or if the study participant declines further treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent.
2. Diagnosis: Histologically or cytologically confirmed diagnosis of cancer which is not amenable to standard therapy, is refractory to standard therapy or for which no standard therapy exists.
3. Age ≥ 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
5. Life expectancy of ≥ 12 weeks.
6. Disease measurability:

   1. Part I (Dose-escalation):

      Participants must have a measurable (as per RECIST criteria version 1.1) and/or evaluable disease (e.g., cytologically or radiologically detectable disease such as ascites, peritoneal deposits, or lesions which do not fulfill RECIST criteria version 1.1 for measurable disease).
   2. Part II (expansion cohort):

   Participants must have at least one measurable disease lesion as per the RECIST criteria version 1.1.
7. Adequate bone marrow function as defined by: WBC of ≥ 3 x109/L, ANC of ≥ 1.5 x 109/L, platelet count of ≥ 100.0 x 109/L, and hemoglobin of ≥ 9g/dL.
8. Adequate liver function, as determined by: Serum total bilirubin ≤1.5 x ULN.AST and ALT ≤ 2.5 x ULN..
9. Adequate renal function assessed by at least one of the following: 1) Serum creatinine ≤ 1.5 x ULN; or 2) creatinine clearance estimate of ≥ 60 mL/min in male and ≥ 50 mL/min in female (as calculated according to Cockcroft-Gault formula).
10. Ability to comply with protocol requirements.
11. Female participants must be postmenopausal (12 months of amenorrhea), surgically sterile or they must agree to use a physical method of contraception. Oral or injectable contraceptive agents cannot be the sole method of contraception. Male participants must be surgically sterile or agree to use a barrier method of contraception.
12. Female participants of child-bearing potential must have a negative serum pregnancy test within the seven days prior to the first IMP administration.

Exclusion Criteria

Participant with any of the following criteria will be excluded from the participation in the study:

1. History of allergic reactions attributed to previous gemcitabine treatment.
2. Symptomatic CNS or leptomeningeal metastases.
3. Prior chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy for bone pain), or immunotherapy within 28 days of first receipt of the IMP (within 6 weeks for nitrosoureas and mitomycin C). Hormone or biological therapy within 14 days of first receipt of IMP.
4. Prior toxicities from chemotherapy or radiotherapy which have not regressed to Grade ≤ 1 severity (NCI-CTCAE version 4.0) apart from neuropathy and alopecia.
5. Another active cancer (excluding basal cell carcinoma or cervical intraepithelial neoplasia (CIN/cervical in situ or melanoma in situ; part II only).
6. Participants with uncontrolled concomitant illness, active infection requiring i.v. antibiotics.
7. Participants will serious illnesses, medical conditions, or other medical history, including laboratory results, which, in the CI or delegates opinion would be likely to interfere with a participant's participation in the study, or with the interpretation of the results.
8. Known HIV or known active Hepatitis B or C.
9. Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc.) that, in the judgment of the CI or delegates may affect the participant's ability to sign the informed consent and undergo study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To determine the RP2D of NUC-1031 administered as either an I.V. weekly or twice-weekly schedule in patients with advanced solid tumours. | 1.5 years
  Adverse events (AE) and changes from baseline in vital signs, clinical laboratory parameters, and electrocardiography (ECG) assessments will be assessed
To further evaluate the safety profile of NUC-1031 in an expanded cohort at RP2D | 1 year
  Adverse events (AE) and changes from baseline in vital signs, clinical laboratory parameters, and electrocardiography (ECG) assessments

SECONDARY OUTCOMES:
To determine the pharmacokinetics of NUC-1031 and its metabolites. | 1.5 years
  PK endpoints will include assessments such as systemic Clearance (CL), Apparent Volume of Distribution (Vd), Area Under the Curve (AUC), Maximum plasma (peak) drug concentration after single dose administration (Cmax), and t1/2.
To explore the preliminary anti-tumour activity of NUC-1031 [given at the RP2D and preferred schedule selected from Part I] | 1 year
  Assessment of anti-tumour activity as defined by RECIST version 1.1
  Urinary excretion of NUC-1031 and metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Blagden, PhD FRCP, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial CRF, London, Hammersmith, United Kingdom